CLINICAL TRIAL: NCT07108842
Title: Evaluation of Postoperative Pain After Using Two Different Irrigation Systems During Endodontic Treatment
Brief Title: Assessment of Pain Using Two Different Irrigation Systems After Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Farhana Altaf, Dr Farhana, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr Farhana
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Pulpal Inflammation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Needle Irrigation (Control Group) (Active Comparator): Patients in this group will receive traditional syringe and needle irrigation during root canal treatment. An open ended irrigation needle will be used to deliver 2.5% sodium hypochlorite into the root canal system. The needle will be placed 1-2 mm short of the working length, and irrigation will be performed intermittently during canal instrumentation. No additional activation method will be used.
  Interventions: Procedure: Conventional Needle Irrigation; Device: Conventional Needle Irrigation (Control Group); Device: Irrigation Solution
- Sonic Irrigation using EndoActivator (Intervention Group) (Experimental): Patients in this group will receive sonic activation of the irrigant using the EndoActivator device during root canal treatment. After instrumentation and irrigation with 2.5% sodium hypochlorite, the irrigant will be activated using the EndoActivator with a medium-sized (25/04) polymer tip. The device will operate at sonic frequencies (~6000 cycles/min) for 30 seconds per canal to enhance irrigant penetration and cleaning efficacy, particularly in the apical third and lateral canals.
  Interventions: Device: endoactivator; Device: Irrigation Solution; Device: Sonic Irrigation with EndoActivator (Experimental Group)

INTERVENTIONS:
Procedure: Conventional Needle Irrigation — Patients in this arm will receive traditional syringe and needle irrigation using a 30-gauge side-vented needle. 2.5% sodium hypochlorite will be used as the irrigant, delivered 1-2 mm short of working length intermittently during root canal instrumentation. No activation device will be used.
  Other Names: Sonic Irrigation with EndoActivator (Experimental Group)
  Arms: Conventional Needle Irrigation (Control Group)
Device: Conventional Needle Irrigation (Control Group) — Patients in this arm will receive traditional syringe and needle irrigation using a 30-gauge side-vented needle. 2.5% sodium hypochlorite will be used as the irrigant, delivered 1-2 mm short of working length intermittently during root canal instrumentation. No activation device will be used.
  Other Names: use of endoactivator
  Arms: Conventional Needle Irrigation (Control Group)
Device: endoactivator — in group 2 irrigation done with endoactivator
  Arms: Sonic Irrigation using EndoActivator (Intervention Group)
Device: Irrigation Solution — irrigation protocol done with disposable syringe
Device: Irrigation Solution — irrigation protocol done with endoactivator
Device: Sonic Irrigation with EndoActivator (Experimental Group) — Patients in this arm will receive sonic activation of the irrigant using the EndoActivator device during root canal treatment. After initial instrumentation and irrigation with 2.5% sodium hypochlorite, the irrigant will be activated using a medium-sized (25/04) EndoActivator tip for 30 seconds per canal at a sonic frequency (~6000 cycles/min), to enhance cleaning and irrigant penetration.
  Arms: Sonic Irrigation using EndoActivator (Intervention Group)

SUMMARY:
assessment of pain using two different irrigation systems after root canal treatment

ELIGIBILITY:
Inclusion Criteria:

1. Single rooted teeth (Anterior or posterior)
2. Teeth with symptomatic irreversible pulpitis with acute apical periodontitis
3. Age group 18-65 years

Exclusion Criteria:

1. Non-restorable teeth, teeth with acute or chronic apical abcess, teeth with internal/external root resorption
2. Teeth with anatomical difficulties like open apices, calcified canals, dilacerations
3. Patients that had any serious medical illness or with systemic disorders
4. Previous root canal treatment
5. Periodontally compromised teeth
6. Presence of sinus tract

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Pain scores will be recorded at 6 hours, 24 hours, and 48 hours after completion of root canal treatment.
  Assessment of postoperative pain intensity using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Analgesic Consumption | 0 to 48 hours after treatment
  Number of analgesic tablets (e.g., ibuprofen/paracetamol) consumed by patients within the first 48 hours post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental hospial, Hitec-IMS, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gondim E Jr, Setzer FC, Dos Carmo CB, Kim S. Postoperative pain after the application of two different irrigation devices in a prospective randomized clinical trial. J Endod. 2010 Aug;36(8):1295-301. doi: 10.1016/j.joen.2010.04.012. Epub 2010 Jun 19. PMID 20647083